CLINICAL TRIAL: NCT00389376
Title: Single and Multiple Dose Escalation Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally Administered Silymarin (Legalon) in Non-Cirrhotic Subjects With Chronic Hepatitis C or Non-Alcoholic Fatty Liver Disease
Brief Title: Phase I Trial of Silymarin for Chronic Liver Diseases
Acronym: SyNCH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: SyNCH Steering Committee, NCCAM/NIDDK/UNC/UPenn/TJU/BIDMC/UPitt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: U01AT003566-01 (NIH); NIH grant # U01-AT0035661
Expanded Access: Available
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Hepatitis C; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Hepatitis C; Non-alcoholic Fatty Liver Disease | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Other): Placebo and 140 mg single dose + every 8 hours
  Interventions: Drug: Placebo; Drug: Silymarin
- Group 2 (Other): Placebo and 280 mg single dose
  Interventions: Drug: Placebo; Drug: Silymarin
- Group 3 (Other): Placebo and 280mg every 8 hours
  Interventions: Drug: Placebo; Drug: Silymarin
- Group 4 (Other): Placebo and 280 single dose + every 8 hours
  Interventions: Drug: Placebo; Drug: Silymarin
- Group 5 (Other): Placebo and 560 mg single dose + every 8 hours
  Interventions: Drug: Placebo; Drug: Silymarin
- Group 6 (Other): Placebo and 560 mg single dose + every 8 hours
  Interventions: Drug: Placebo; Drug: Silymarin
- Group 7 (Other): Placebo and 700 mg single dose + every 8 hours
  Interventions: Drug: Placebo; Drug: Silymarin

INTERVENTIONS:
Drug: Placebo — Placebo
Drug: Silymarin — 140 mg every 8 hours
  Other Names: Legalon
  Arms: Group 1
Drug: Silymarin — 280 mg single dose
  Other Names: Legalon
  Arms: Group 2
Drug: Silymarin — 280 mg single dose + every 8 hours
  Other Names: Legalon
  Arms: Group 4
Drug: Silymarin — 560 mg single dose + every 8 hours
  Other Names: Legalon
  Arms: Group 5
Drug: Silymarin — 560 mg single dose + every 8 hours
  Other Names: Legalon
  Arms: Group 6
Drug: Silymarin — 280 mg every 8 hours
  Other Names: Legalon
  Arms: Group 3
Drug: Silymarin — 700 mg single dose + every 8 hours
  Other Names: Legalon
  Arms: Group 7

SUMMARY:
The purpose of this study is to determine the safety and tolerability of different dosages of silymarin on subjects with Hepatitis C or Non-Alcoholic Fatty Liver Disease.

ELIGIBILITY:
Inclusion criteria

Subjects will be eligible for enrollment in this study if they meet the following criteria:

* Males or females; age at least 18 years at screening
* Abnormal ALT > 65 IU/L (ie, approximately 1.5 x upper limit of normal)
* Negative urine pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of silymarin. Females of childbearing potential must be using two reliable forms of effective contraception during the study (while on drug and during follow-up)
* Hepatitis C virus (HCV) patients
* Previous treatment with any interferon-based therapy without sustained virological response.
* Serum HCV RNA above quantifiable level of detection by the assay, within 1 year of screening and after the end of therapy
* No antiviral therapy for at least 6 months prior to screening visit
* Nonalcoholic fatty liver disease (NAFLD) patients:
* Liver biopsy compatible with NAFLD within 3 years of screening
* Absence of other liver diseases by serological screening (anti-HCV, HBsAg), historical serological data from within 3 years of screening is acceptable.
* Before entering the study, subjects must agree not to consume alcohol for 48 hours prior to PK sampling days or while on study.

Exclusion criteria

Subjects with any of the following will not be eligible for participation:

* Use of silymarin or other milk thistle preparations within 30 days of screening
* Use of other antioxidants such as vitamin E, vitamin C, glutathione, alpha-tocopherol, within 30 days of screening. A multivitamin at standard doses will be allowed.
* Allergy/sensitivity to milk thistle or its preparations
* Use of silymarin or other antioxidants (as above) during the screening period.
* Use of warfarin, metronidazole or chronic use of acetaminophen greater than two gram per day
* Previous liver biopsy that demonstrated presence of cirrhosis
* Previous liver biopsy that demonstrated greater than or equal to 15% steatosis or evidence of steatohepatitis for HCV cohort
* Positive test for anti-HIV or HBsAg within 3 years of screening
* Positive urine drug screen for drugs of abuse at screening
* Alcohol consumption of more than one drink or equivalent (>12 grams) per day. Patients who consumed more than this in the past must have maintained a level 12 grams or less per day of alcohol consumption for at least six months prior to screening.
* History of other chronic liver disease, including metabolic diseases, documented by appropriate test(s)
* Women with ongoing pregnancy or breast-feeding, or contemplating pregnancy
* Platelet count <130,000 cells/mm3.
* Serum creatinine level >1.5 times the upper limit of normal at screening, or CrCl 60 cc/min, or currently on dialysis. The creatinine clearance (CrCl) will be calculated according to Cockcroft-Gault.
* Evidence of alcohol or drug abuse within 6 months prior to screening
* Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dl, total bilirubin > 1.5 mg/dl, or PT/INR > 1.3 times normal at screening, or history or presence of ascites or encephalopathy, or bleeding from esophageal varices
* History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, or active gastrointestinal conditions that might interfere with drug absorption)
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hepatitis, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis) that could affect inflammatory biomarkers
* History of solid organ or bone marrow transplantation
* History of thyroid disease poorly controlled on prescribed medications
* Use of oral steroids within 30 days prior to screening
* Concurrent medications that are CYP3A4 inducers
* Inability or unwillingness to provide informed consent or abide by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: K. Rajender Reddy, MD, Principal Investigator — University of Pennsylvania; Victor Navarro, MD, Principal Investigator — Thomas Jefferson University; Nezam Afdhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Michael Fried, MD, Principal Investigator — University of North Carolina
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Graduate School of Public Health, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Schrieber SJ, Hawke RL, Wen Z, Smith PC, Reddy KR, Wahed AS, Belle SH, Afdhal NH, Navarro VJ, Meyers CM, Doo E, Fried MW. Differences in the disposition of silymarin between patients with nonalcoholic fatty liver disease and chronic hepatitis C. Drug Metab Dispos. 2011 Dec;39(12):2182-90. doi: 10.1124/dmd.111.040212. Epub 2011 Aug 24. PMID 21865319